CLINICAL TRIAL: NCT04487600
Title: A Randomized, Controlled Trial Comparing Active vs. Passive Voiding Trials in a Gynecologic Oncologic Patient Population Undergoing Same-day Discharge Hysterectomy
Brief Title: The Impact of Post-operative Voiding Trial on Length of Stay Following Laparoscopic Hysterectomy: A Prospective, Randomized Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Colleen Marie Feltmate, MD, BWPO Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2015P000902
Record Dates: First submitted 2020-07-17; First posted 2020-07-27 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Minimally Invasive Surgical Procedure; Hysterectomy; Urinary Retention
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Intervention Model Description: Patients who were scheduled to undergo a same day discharge laparoscopic hysterectomy were assessed for eligibility to participate in this study. A computer generated blocked randomization schema was utilized with alternating block sizes to determine study groups. Participants were randomized 1:1 to each study group (active voiding trial vs. passive voiding trial). There was no cross-over between arms. If the participant did not receive the study intervention as allocated they were withdrawn from the study.
Who Masked: Investigator
Masking Description: Voiding trial protocols for each group (AVT and PVT) as well as data collection sheets were stored in sequentially numbered, opaque, sealed envelopes which were assigned after enrollment and were opened in the operating room at the completion of surgery by the surgical assistant. Attending surgeons and investigators were blinded to the individual patient study assignment. Due to the nature of the study, participants were not masked to their intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Voiding Trial (Experimental): At the completion of surgery, a Foley catheter was left in place. When the patient was determined to be ambulatory by the recovery room nurse, the bladder was backfilled with 300cc of sterile normal saline. Voiding 200cc or (2/3) of the backfill amount was considered passing.
  Interventions: Other: Active voiding trial
- Passive Voiding Trial (No Intervention): At the completion of surgery, a Foley catheter was removed in the operating room. Study participants were allowed six hours to void spontaneously, with 200cc being considered adequate consistent with institution standard practice. At the completion of six hours, if spontaneous voiding has not occurred, a bladder scan was performed and additional time was allowed based on bladder volume with criteria previously established as institution standards based on published practices.

INTERVENTIONS:
Other: Active voiding trial
  Arms: Active Voiding Trial

SUMMARY:
The aim of this study is to investigate the impact of an active voiding trial compared to a passive voiding trial on time to discharge following a planned same day discharge laparoscopic hysterectomy. The investigators hypothesize that performing an active voiding trial will assess urinary function and lead to a reduction in length of stay.

DETAILED DESCRIPTION:
Following laparoscopic surgery with hysterectomy, there is no standard method for assuring urinary function prior to discharge. Total laparoscopic hysterectomy (TLH) has been demonstrated to be safe with a reduction in post-operative morbidity and length of hospital stay with no difference in cancer related outcomes in endometrial cancer. Furthermore, the investigators have demonstrated that following the adoption of same day discharge, there was no difference in composite complication rates or readmissions. Awaiting a passive void trial may impact time to discharge as well as same day discharge; however, this has not been clearly studied in this patient population. The aim of this study is to determine the difference in time to discharge following an active voiding trial with bladder backfill in the post-operative recovery unit compared to a passive voiding trial with removal of the Foley catheter in the operating room at the end of the procedure. Secondary outcomes include time to void, catheter replacement, discomfort with the voiding trial, and overnight admission.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo a total laparoscopic hysterectomy by a gynecologic oncology surgeon for either benign or malignant disease
* planned same day discharge surgery

Exclusion Criteria:

* history of significant urinary dysfunction (such as home catheterization) or neurologic dysfunction precluding spontaneous voiding
* bilateral radical pelvic dissection (defined as bilateral ureterolysis or removal of bilateral parametria)
* surgical cases converted to laparotomy or open surgery
* Surgical or medical contra-indications (based on the surgeons or anesthesiologists' recommendations) to same day discharge requiring inpatient admission

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Given the nature of the surgery (gynecologic oncology surgery with hysterectomy) the study is limited to female participants
Enrollment: 130 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-08-04 (Actual); Study Completion 2017-08-04 (Actual)

PRIMARY OUTCOMES:
length of hospital stay | within 24 hours (1440 minutes) following surgical procedure (while most participants are discharged on the same day some participants require overnight admission with length of stay up to 24 hours- though still measured in minutes)
  Time (minutes) from the completion of surgery to discharge from the post-operative recovery unit

SECONDARY OUTCOMES:
time to void | within 12 hours (720 minutes) following surgical procedure
  Time (minutes) from Foley catheter removal to adequate voiding
catheter replacement | within 24 hours (1440 minutes) following surgical procedure
  failed trial of void (unable to void adequate volume 2/3rd of backfill or 200cc) requiring replacement of a Foley catheter for post-operative urinary retention
discomfort with voiding trial | within 12 hours (720 minutes) following surgical procedure
  average pain scale as measured by Wong-Baker FACES Pain Rating Scale ranging from 0 to 10 with 0 being no pain and 10 being the worst pain.
overnight admission | within 1 day following surgical procedure
  planned same day discharge requiring an unplanned admission to the extended recovery unit (ERU)

IPD SHARING:
Plan to Share IPD: Yes
De-identified patient data and voiding protocols will be made available upon request via email to other researchers
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available upon request until the time of publication.
Access Criteria: requests should be made via the study contact email.

REFERENCES:
- [Background] Lee J, Jennings K, Borahay MA, Rodriguez AM, Kilic GS, Snyder RR, Patel PR. Trends in the national distribution of laparoscopic hysterectomies from 2003 to 2010. J Minim Invasive Gynecol. 2014 Jul-Aug;21(4):656-61. doi: 10.1016/j.jmig.2014.01.012. Epub 2014 Jan 24. PMID 24462854
- [Background] Pitter MC, Simmonds C, Seshadri-Kreaden U, Hubert HB. The impact of different surgical modalities for hysterectomy on satisfaction and patient reported outcomes. Interact J Med Res. 2014 Jul 17;3(3):e11. doi: 10.2196/ijmr.3160. PMID 25048103
- [Background] Schiavone MB, Herzog TJ, Ananth CV, Wilde ET, Lewin SN, Burke WM, Lu YS, Neugut AI, Hershman DL, Wright JD. Feasibility and economic impact of same-day discharge for women who undergo laparoscopic hysterectomy. Am J Obstet Gynecol. 2012 Nov;207(5):382.e1-9. doi: 10.1016/j.ajog.2012.09.014. Epub 2012 Sep 17. PMID 23107080
- [Background] Walker JL, Piedmonte MR, Spirtos NM, Eisenkop SM, Schlaerth JB, Mannel RS, Spiegel G, Barakat R, Pearl ML, Sharma SK. Laparoscopy compared with laparotomy for comprehensive surgical staging of uterine cancer: Gynecologic Oncology Group Study LAP2. J Clin Oncol. 2009 Nov 10;27(32):5331-6. doi: 10.1200/JCO.2009.22.3248. Epub 2009 Oct 5. PMID 19805679
- [Background] Walker JL, Piedmonte MR, Spirtos NM, Eisenkop SM, Schlaerth JB, Mannel RS, Barakat R, Pearl ML, Sharma SK. Recurrence and survival after random assignment to laparoscopy versus laparotomy for comprehensive surgical staging of uterine cancer: Gynecologic Oncology Group LAP2 Study. J Clin Oncol. 2012 Mar 1;30(7):695-700. doi: 10.1200/JCO.2011.38.8645. Epub 2012 Jan 30. PMID 22291074
- [Background] Melamed A, Katz Eriksen JL, Hinchcliff EM, Worley MJ Jr, Berkowitz RS, Horowitz NS, Muto MG, Urman RD, Feltmate CM. Same-Day Discharge After Laparoscopic Hysterectomy for Endometrial Cancer. Ann Surg Oncol. 2016 Jan;23(1):178-85. doi: 10.1245/s10434-015-4582-4. Epub 2015 May 9. PMID 25956576
- [Background] Nahas S, Feigenberg T, Park S. Feasibility and safety of same-day discharge after minimally invasive hysterectomy in gynecologic oncology: A systematic review of the literature. Gynecol Oncol. 2016 Nov;143(2):439-442. doi: 10.1016/j.ygyno.2016.07.113. Epub 2016 Jul 27. PMID 27475523
- [Background] Geller EJ. Prevention and management of postoperative urinary retention after urogynecologic surgery. Int J Womens Health. 2014 Aug 28;6:829-38. doi: 10.2147/IJWH.S55383. eCollection 2014. PMID 25210477
- [Background] Foundation W-BF. Wong-Baker FACES® Pain Rating Scale. 2016
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Result] Ghezzi F, Cromi A, Uccella S, Colombo G, Salvatore S, Tomera S, Bolis P. Immediate Foley removal after laparoscopic and vaginal hysterectomy: determinants of postoperative urinary retention. J Minim Invasive Gynecol. 2007 Nov-Dec;14(6):706-11. doi: 10.1016/j.jmig.2007.06.013. PMID 17980330
- [Result] Geller EJ, Hankins KJ, Parnell BA, Robinson BL, Dunivan GC. Diagnostic accuracy of retrograde and spontaneous voiding trials for postoperative voiding dysfunction: a randomized controlled trial. Obstet Gynecol. 2011 Sep;118(3):637-642. doi: 10.1097/AOG.0b013e318229e8dd. PMID 21860294
- [Result] Foster RT Sr, Borawski KM, South MM, Weidner AC, Webster GD, Amundsen CL. A randomized, controlled trial evaluating 2 techniques of postoperative bladder testing after transvaginal surgery. Am J Obstet Gynecol. 2007 Dec;197(6):627.e1-4. doi: 10.1016/j.ajog.2007.08.017. PMID 18060956
- [Result] Pulvino JQ, Duecy EE, Buchsbaum GM, Flynn MK. Comparison of 2 techniques to predict voiding efficiency after inpatient urogynecologic surgery. J Urol. 2010 Oct;184(4):1408-12. doi: 10.1016/j.juro.2010.05.096. Epub 2010 Aug 19. PMID 20727543
- [Result] Alessandri F, Mistrangelo E, Lijoi D, Ferrero S, Ragni N. A prospective, randomized trial comparing immediate versus delayed catheter removal following hysterectomy. Acta Obstet Gynecol Scand. 2006;85(6):716-20. doi: 10.1080/00016340600606976. PMID 16752265